CLINICAL TRIAL: NCT05269524
Title: TAILORED INTERNET-DELIVERED COGNTIVE BEHAVIOR THERAPY FOR DEPRESSED OLDER ADULTS: A RANDOMIZED TRIAL
Brief Title: ICBT for Depression in Older Adults
Acronym: ALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alm study
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Internet Treatment; Active Control
Keywords: depression; Internet-delivered cognitive-behavior therapy; Older adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Therapist-guided internet treatment.
  Interventions: Behavioral: Internet-delivered tailored cognitive behavior therapy
- Attention control (Active Comparator): Non-directive supportive contact via email.
  Interventions: Behavioral: Internet-delivered tailored cognitive behavior therapy

INTERVENTIONS:
Behavioral: Internet-delivered tailored cognitive behavior therapy — Therapists-supported tailored 10-week treatment for depression in older adults.
  Other Names: ICBT

SUMMARY:
The study was a randomized controlled trial investigating treatment effects against an active control condition. 101 self-recruited participants, aged 65 to 88 years, were included. The intervention was a 10-week internet-based tailored CBT protocol consisting of 6-10 pre-defined modules tailored to patient profile and preferences. Participants in the treatment group benefitted more than participants in the control condition on almost all measures with moderate between-group effect-sizes.

DETAILED DESCRIPTION:
Depression in older adults is associated with poorer functioning, worsened cognitive impairment and disability, as well as medical illnesses. It can also increase the risk of suicide and is associated with a high usage of medical services. It is common that depressive symptoms co-occur with other psychiatric symptoms (i.e. anxiety). In the case of co-morbidity, patients present with greater difficulties and the problems tend to be more persistent. Together this stresses the importance of developing effective treatments. Psychological treatments can be effective but are rarely offered and thus alternative modes of treatment delivery should be considered such as internet interventions. Design: The study was a randomized controlled trial investigating treatment effects against an active control condition. Participants: 101 self-recruited participants, aged 65 to 88 years, were included. Intervention: The intervention was a 10-week internet-based tailored CBT protocol consisting of 6-10 pre-defined modules tailored to patient profile and preferences. Measurements: Depression, anxiety, life quality and cognitive decline were assessed through self-reported measures together with an online test of cognitive flexibility. Results: Participants in the treatment group benefitted more than participants in the control condition on almost all measures with moderate between-group effect-sizes. Cognitive decline improved during treatment and neither cognitive decline, nor cognitive flexibility predicted treatment outcome. Conclusion: The study adds to the evidence of internet-delivered psychological treatment for depression, with or without psychiatric comorbidities, in older adults. It also highlights the possibility of perceived cognitive decline as being part of the clinical picture and reversible, rather than reason for exclusion from for psychological treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* presence of depressive symptoms
* living in Sweden
* access to the internet and a computer on a regular basis.

Exclusion Criteria:

* heightened suicidal ideation
* drug or alcohol abuse or dependency
* other ongoing psychological treatment
* severe psychiatric or cognitive problems
* unstable psychopharmacological medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale (GDS) | Change pre to 10-week post
  GDS scores range between 0 and 15, and five or less are considered within normal range

SECONDARY OUTCOMES:
Beck Depression Inventory II | Change pre to 10-week post
  For the 21 item BDI-II the maximum score is 63 points and scores below 14 are considered minimal depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
On request and in collaboration.

REFERENCES:
- [Derived] Nordgren LB, Ludvigsson M, Silfvernagel K, Tornhage L, Savas L, Soderqvist S, Dinnetz S, Henrichsen P, Larsson J, Strom H, Lindh M, Berger T, Andersson G. Tailored internet-delivered cognitive behavior therapy for depression in older adults: a randomized controlled trial. BMC Geriatr. 2024 Dec 10;24(1):998. doi: 10.1186/s12877-024-05597-8. PMID 39658784